CLINICAL TRIAL: NCT01668836
Title: Influence of Caloric Restriction and Resveratrol in the Sirtuin System in Women and Men Aged 55 to 65 Years.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, ANTONIO DE PADUA MANSUR, PHD, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 788012; 2012/01051-5 (Other Grant/Funding Number: FAPESP - SAO PAULO RESEARCH FOUNDATION)
Record Dates: First submitted 2012-08-14; First posted 2012-08-20 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Vascular System Injuries; Lipid Metabolism Disorders; Endothelial Disfunction
Keywords: sirtuin; atherosclerosis; longevity; calorie restriction; resveratrol; vascular reactivity
MeSH Terms: conditions — Vascular System Injuries; Lipid Metabolism Disorders; Atherosclerosis | interventions — Resveratrol; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- men with resveratrol (Experimental): 12 men will receive a pill with 500mg of resveratrol daily for 30 days
  Interventions: Drug: Resveratrol
- women with resveratrol (Experimental): 12 women will receive a pill with 500mg of resveratrol daily for 30 days
  Interventions: Drug: Resveratrol
- men with caloric restriction (Active Comparator): 12 men will follow a 1000 calories per day diet for 30 days
  Interventions: Behavioral: Caloric restriction
- women with caloric restriction (Active Comparator): 12 women will follow a 1000 calories per day diet for 30 days
  Interventions: Behavioral: Caloric restriction

INTERVENTIONS:
Drug: Resveratrol — 1 pill daily containing 500 mg/d of resveratrol for 30 days
  Arms: men with resveratrol; women with resveratrol
Behavioral: Caloric restriction — Diet of 1000kcal per day for 30 days
  Arms: men with caloric restriction; women with caloric restriction

SUMMARY:
Women have a natural protection that gives them greater longevity. One hypothesis most commonly used is the estrogen protection in the premenopausal period. However many studies of various forms of hormone replacement therapy proved ineffective in promoting additional protection for women. Thus, it is discussed other ways of protection associated with longevity in women. Of these, the sirtuin system was found in several animal studies to be associated with longevity. This system also showed, through the involvement of several metabolic pathways, an important protection against the process of atherosclerosis. But the activity of this system in humans is unknown and if it is more active in women than in men. The study's main objectives are to analyze this system in healthy 24 women and 24 men aged 55 to 65 years, and their influence on the main metabolic pathways related to longevity and the process of atherosclerosis. The research protocol includes analysis of the influence of sirtuin (SIRT1) in vascular reactivity, lipid profile, antioxidant capacity, markers of inflammation and homeostasis, before and after the interventions with caloric restriction or resveratrol administration. It is expected of this study mechanistic conclusion for longevity and possible clinical applications in the mechanism of atherosclerosis prevention.

DETAILED DESCRIPTION:
After a washout period of 15 days without medication, men and women will be randomized to the group of calorie restriction or resveratrol so that in 24 individuals (12 women and 12 men) will be given a hypocaloric diet (1000 calories per day) and the remaining 24 individuals (12 women and 12 men), a daily pill of 500mg of resveratrol. In the two moments, after the washout period and before the intervention (baseline) and after 30 days of intervention (final) will evaluate the clinical, laboratory and vascular reactivity of all subjects.

ELIGIBILITY:
Inclusion Criteria:

* clinical history, physical examination and electrocardiogram normal

Exclusion Criteria:

* premenopausal women (less than 1 year of natural amenorrhea)
* Body mass index ≥ 35 kg/m2
* Smoking
* Severe hypertension (diastolic blood pressure ≥ 110 mmHg)
* Severe dyslipidemia (triglycerides ≥ 500mg/dL, total cholesterol ≥ 300mg/dL)
* Diabetes
* Previous using previous statins or hormone replacement therapy. Other exclusion criteria are: chronic renal failure (serum creatinine ≥ 2.0 mg / dl), hepatic, endocrine, hematologic, respiratory or metabolic clinically significant.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antônio de Pádua Mansur, PHD, Principal Investigator — InCor Heart Institute
Locations (1):
- INCOR - Heart Institute, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Men With Caloric Restriction: 12 men will follow a 1000kcal/day diet for 30 days
  Caloric restriction: Diet of 1000kcal per day for 30 days
- Women With Caloric Restriction: 12 women will follow a 1000kcal/day diet for 30 days
  Caloric restriction: Diet of 1000kcal per day for 30 days
Period: Overall Study
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Men With Caloric Restriction: 12 men will follow a 1000kcal/day diet for 30 days
  Caloric restriction: Diet of 1,000kcal per day for 30 days
- Women With Caloric Restriction: 12 women will follow a 1000kcal/day diet for 30 days
  Caloric restriction: Diet of 1,000kcal per day for 30 days
- Total: Total of all reporting groups
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (3.6) | 58.5 (3.4) | 57.7 (3.5) | 59.5 (3.7) | 58.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 12 | 0 | 12 | 24
  Male | 12 | 0 | 12 | 0 | 24
Region of Enrollment [Number; unit: participants]
  Brazil | 12 | 12 | 12 | 12 | 48
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] | 28.5 (4.4) | 26.5 (3.4) | 26.2 (3.5) | 25.5 (3.7) | 26.7 (3.8)
abdominal circumference [Mean (Standard Deviation); unit: cm] | 100.9 (13.9) | 92.7 (8.7) | 96.5 (7.6) | 92 (7) | 95.5 (10)
heart rate [Mean (Standard Deviation); unit: beats/minute] | 63.6 (7.9) | 65.6 (9.1) | 63.9 (10.7) | 60.8 (8.3) | 63.6 (9.0)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 136.9 (15.0) | 126 (14.5) | 133.2 (16.6) | 125.6 (14.1) | 130.6 (15.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 83.9 (12.0) | 78.5 (9.3) | 84.8 (9.9) | 80.6 (12.3) | 82 (10.8)
total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 192.8 (28.1) | 222.7 (32.5) | 197.3 (36.2) | 235.1 (44.9) | 212.0 (39.1)
HDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 43.6 (10.2) | 54.8 (15.2) | 43.5 (9.0) | 67.2 (18.2) | 52.3 (16.5)
LDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 125.5 (29.9) | 140.8 (28.7) | 127.6 (34.0) | 149.8 (37.6) | 135.5 (32.0)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 126.5 (63.0) | 121.6 (72.4) | 131.0 (77.9) | 91.4 (37.4) | 117.6 (64.4)
C-reactive protein [Mean (Standard Deviation); unit: mg/dL] | 1.13 (0.67) | 3.47 (2.38) | 1.63 (1.01) | 2.31 (2.44) | 2.13 (1.92)
Apolipoprotein A1 [Mean (Standard Deviation); unit: g/L] | 1.37 (0.21) | 1.53 (0.19) | 1.34 (0.11) | 1.72 (0.25) | 1.49 (0.24)
Apolipoprotein B [Mean (Standard Deviation); unit: g/L] | 0.91 (0.18) | 1.04 (0.28) | 0.97 (0.25) | 1.04 (0.27) | 0.99 (0.25)
lipoprotein (a) [Mean (Standard Deviation); unit: mg/dL] | 16.2 (20.1) | 24.1 (29.7) | 31.8 (44.7) | 23.9 (17.4) | 24.0 (29.5)
glucose [Mean (Standard Deviation); unit: mg/dL] | 95.8 (14.1) | 96.3 (13.8) | 91.8 (12.6) | 95.4 (8.5) | 94.8 (12.2)
luteinizing hormone [Mean (Standard Deviation); unit: microUI/mL] | 3.34 (1.67) | 20.9 (7.53) | 4.46 (1.95) | 29.9 (9.05) | 14.7 (12.7)
follicle stimulating hormone [Mean (Standard Deviation); unit: microUI/mL] | 4.12 (2.2) | 60.8 (20.4) | 6.22 (3.53) | 75.8 (18.7) | 36.8 (35.1)
Estradiol [Mean (Standard Deviation); unit: pg/mL] | 36.4 (10.5) | 38.6 (16.4) | 43.4 (12.3) | 25.9 (8.3) | 36.0 (13.5)
norepinephrine [Mean (Standard Deviation); unit: pg/mL] | 267.8 (148.9) | 270.8 (88.6) | 286.3 (126.8) | 420.9 (171.0) | 306.7 (144.5)
Insulin [Mean (Standard Deviation); unit: microUI/L] | 53.7 (33.7) | 77.1 (62.2) | 69.3 (57.1) | 44.3 (28.9) | 61.5 (48.2)
Sirtuin [Mean (Standard Deviation); unit: ng/mL] | 0.95 (0.46) | 1.16 (0.90) | 1.65 (1.40) | 1.65 (2.21) | 1.35 (1.39)
Estrone [Mean (Standard Deviation); unit: pg/mL] | 17.6 (18.3) | 12.4 (17.4) | 3.1 (0.0) | 5.11 (6.7) | 10.0 (14.7)
Sirtuin-1 gene expression by real time polimerase chain reaction "RT-PCR" [Mean (Standard Deviation); unit: arbitrary unit] — Values obtained from delta CT (cycle threshold) using as normalizer GAPDH gene.
  arbitrary unit | 10.4 (1.28) | 11.6 (1.38) | 11.4 (1.26) | 10.6 (1.15) | 11.0 (1.33)
RAGE (receptor for advanced glycation end-products) gene expression "RT-PCR" [Mean (Standard Deviation); unit: arbitrary unit] | 11.3 (1.24) | 12.7 (1.65) | 10.9 (1.68) | 10.5 (1.76) | 11.3 (1.74)
Platelet aggregation by adenosine diphosphate (ADP) [Mean (Standard Deviation); unit: %] — percentage of maximum amplitude aggregation by adenosine diphosphate
  % | 86.13 (4.06) | 88.90 (5.87) | 84.20 (7.80) | 88.45 (3.65) | 86.92 (5.74)
Platelet aggregation by epinephrine [Mean (Standard Deviation); unit: %] — percentage of maximum amplitude aggregation
  % | 84.23 (3.90) | 83.42 (10.22) | 66.88 (25.92) | 81.20 (18.27) | 78.93 (17.72)
Nonesterified fatty acid [Mean (Standard Deviation); unit: mmol/L] | 25.73 (16.55) | 18.64 (14.12) | 29.75 (49.34) | 24.17 (20.92) | 24.67 (28.69)
Clot onset time [Mean (Standard Deviation); unit: seconds] | 38.25 (4.16) | 30.75 (9.58) | 38.25 (4.00) | 91.64 (177.95) | 48.83 (86.58)
Clot complete [Mean (Standard Deviation); unit: seconds] | 103.83 (13.67) | 80.83 (12.01) | 100.17 (14.32) | 152.64 (211.01) | 108.45 (102.45)
Slope [Mean (Standard Deviation); unit: Pascal/min] — Slope reflects activity of fibrinogen and platelet function. Denotes the speed at which solid clot was formed. Its value is reduced in presence of low levels of fibrinogen and platelet function. It shows the strength which the clot is formed.
  Pascal/min | 100.83 (38.42) | 165.42 (60.43) | 108.17 (43.98) | 158.36 (37.85) | 132.66 (53.47)
Max Elasticity [Mean (Standard Deviation); unit: Pascal] | 1598.50 (398.18) | 2202.98 (391.50) | 1639.82 (383.97) | 2164.64 (275.91) | 1895.88 (456.53)

OUTCOME MEASURES:

1. Primary Outcome: Direct Evaluation of the Sirtuin 1 Gene Expression
Description: The Sirtuin 1 gene expression was measured by real time PCR in peripheric blood. Unit of measure was arbitrary unit. "Arbitrary unit was relative to the control gene expression (control gene = 1)".
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: arbitrary unit relative to control gene
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
arbitrary unit relative to control gene | 11.04 (1.75) | 11.43 (1.42) | 12.84 (1.36) | 12.05 (1.13)

2. Secondary Outcome: Influence of the Sirtuin 1 System on Lipid Profile, Glucose, and C-reactive Protein.
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  - serum HDL, LDL, lipoprotein(a), C reactive protein, glucose.
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "mg/dL"
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"mg/dL"
  HDL-cholesterol "mg/dL" | 43.00 (10.37) | 53.33 (15.11) | 41.08 (9.10) | 62.92 (15.16)
  LDL-cholesterol "mg/dL" | 125.50 (29.93) | 153.58 (45.92) | 126.33 (33.47) | 134.25 (34.27)
  Lipoprotein(a)"mg/dL" | 15.03 (19.98) | 24.43 (33.57) | 32.73 (41.34) | 20.86 (12.82)
  total cholesterol "mg/dL" | 196.08 (31.67) | 239.08 (47.12) | 193.83 (37.20) | 211.50 (41.79)
  Triglycerides "mg/dL" | 137.75 (62.22) | 159.50 (118.13) | 131.00 (77.91) | 72.25 (30.58)
  C-reactive protein "mg/dL" | 0.13 (0.14) | 0.28 (0.23) | 0.17 (0.14) | 0.16 (0.11)
  glucose "mg/dL" | 99.83 (16.29) | 97.33 (12.51) | 89.92 (5.78) | 91.17 (6.19)

3. Other Pre Specified Outcome: Differences Between Men and Women.
Description: We will also compare women vs men baseline and final data.
Time Frame: 30 days
Reporting Status: Not Posted

4. Primary Outcome: Sirtuin
Description: Sirtuin plasma levels before and 30 days post-treatment
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL | 4.84 (2.78) | 6.67 (2.99) | 6.14 (1.98) | 5.46 (2.51)

5. Secondary Outcome: Influence of the Sirtuin 1 System on Apolipoproteins AI and B.
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  - apolipoproteins AI and B
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "g/dL"
Groups:
- Men With Resveratrol: 12 men will receive a pill with 500mg of resveratrol
- Women With Resveratrol: 12 women will receive a pill with 500mg of resveratrol
- Men With Caloric Restriction: 12 men will follow a 1000Kcal/day of caloric restriction
- Women With Caloric Restriction: 12 women will follow a 1000Kcal/day of caloric restriction
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"g/dL"
  Apolipoprotein A1 "g/dL" | 1.33 (0.20) | 1.55 (0.24) | 1.29 (0.21) | 1.57 (0.29)
  Apolipoprotein B "g/dL" | 0.95 (0.19) | 1.13 (0.31) | 0.97 (0.27) | 0.93 (0.26)

6. Secondary Outcome: Influence of the Sirtuin 1 System on Estradiol
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  - estradiol
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "pg/mL"
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"pg/mL" | 38.92 (13.60) | 34.81 (12.73) | 42.13 (14.26) | 29.05 (7.67)

7. Secondary Outcome: Influence of the Sirtuin 1 System on Platelet Aggregation.
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  - platelet aggregation by ADP and norepinephrine.
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: percentage platelet aggregation
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage platelet aggregation
  Platelet aggregation by ADP "%" | 88.03 (4.92) | 88.96 (4.15) | 87.32 (4.12) | 87.24 (12.06)
  Platelet aggregation by norepinephrine "%" | 81.06 (10.46) | 81.77 (16.91) | 74.43 (23.83) | 72.09 (27.37)

8. Secondary Outcome: Influence of the Sirtuin 1 System on Biomarkers
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  - non-esterified fatty acids, insulin, luteinizing hormone, follicle stimulating hormone.
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "microUI/mL"
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"microUI/mL"
  Non sterified fatty acid "microUI/mL" | 22.45 (10.32) | 23.73 (12.51) | 8.83 (8.73) | 24.67 (19.43)
  Insulin "microUI/mL" | 79.00 (54.55) | 80.58 (64.15) | 53.25 (32.28) | 67.08 (30.20)
  Luteinizing hormone "microUI/mL" | 3.93 (1.66) | 19.97 (7.01) | 4.50 (1.65) | 28.56 (11.77)
  Follicle stimulating hormone "microUI/mL" | 4.40 (2.26) | 57.78 (15.35) | 6.31 (3.71) | 79.79 (26.04)

9. Secondary Outcome: Influence of the Sirtuin 1 System on Estrone and Norepinephrine.
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  - estrone, norepinephrine.
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "pg/dL"
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"pg/dL"
  Norepinephrine "pg/dL" | 219.33 (99.24) | 227.83 (92.13) | 190.83 (124.82) | 329.00 (194.11)
  Estrone"pg/dL" | 14.92 (18.54) | 13.23 (15.49) | 7.62 (15.68) | 4.12 (3.52)

10. Secondary Outcome: Influence of the Sirtuin 1 System on Receptor for Advanced Glycation End Products (RAGE) Gene Expression
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  * RAGE gene expression
  * "Arbitrary unit was relative to the control gene expression (control gene = 1)"
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: arbitrary unit relative to control gene
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
arbitrary unit relative to control gene | 11.88 (1.80) | 12.78 (1.38) | 12.17 (1.99) | 11.75 (1.74)

11. Secondary Outcome: Influence of the Sirtuin 1 System on Thromboelastography Clot Formation.
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  -dynamics of clot formation: clot onset time and clot complet
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "sec"
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"sec"
  Clot onset time "sec" | 38.00 (5.62) | 35.50 (5.50) | 40.42 (7.93) | 35.67 (5.82)
  Clot complet "sec" | 100.83 (17.47) | 89.00 (16.59) | 101.00 (23.68) | 86.83 (15.75)

12. Secondary Outcome: Influence of the Sirtuin 1 System on Thromboelastography.
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  - slope of clot formation dynamics
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "Pascal/min"
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"Pascal/min" | 106.83 (50.13) | 158.67 (47.13) | 115.42 (67.38) | 156.75 (43.42)

13. Secondary Outcome: Influence of the Sirtuin 1 System on Max Elasticity of Clot on Thromboelastography.
Description: For indirect analysis of the sirtuin 1 system, the following procedures will be done before and after the intervention with caloric restriction or resveratrol administration:
  -max elasticity of clot on thromboelastography
Time Frame: 30 days post-treatment
Measure: Mean (Standard Deviation); unit: "Pascal"
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Number analyzed (Participants) | 12 | 12 | 12 | 12
"Pascal" | 1690.58 (522.54) | 2059.83 (337.48) | 1691.50 (380.49) | 2041.12 (318.71)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Men With Resveratrol | Women With Resveratrol | Men With Caloric Restriction | Women With Caloric Restriction
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No